CLINICAL TRIAL: NCT03555227
Title: Ultrasound Guided (USG) PECS Versus Local Infiltration Anaesthesia (LIA) for Breast Cancer Surgery - A Randomized Quadruple Blinded Efficacy and Safety Study
Brief Title: USG PECS vs LIA for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Service, United Kingdom (Other Government)
Collaborators: Southern Health and Social Care Trust (Other Government)
Responsible Party: Principal Investigator, Shiva ARAVA, Doctor, Consultant Anaesthetist, National Health Service, United Kingdom
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST1516/35-193503
Record Dates: First submitted 2018-05-18; First posted 2018-06-13 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer Female
Keywords: breast cancer analgesia; pecs2 blocks; ultrasound
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a single-centre, prospective; double blinded randomised case control interventional study.Patients will be randomly allocated to group X or Y. Following anesthesia induction, all patients will receive USG modified Pecs2 blocks as described by Blanco et al with 30 mls of pharmacy prepared Drug A (active drug 0.25% levobupivacaine) or Drug P (placebo 0.9% NaCl), labelled "PRE" respectively based on the group allocation. After surgery, the surgeon shall infiltrate the wound with 30 mls of Drug P or Drug A respectively, labelled "POST". Drug P has no active role in terms of outcomes being assessed in this study. Intraoperative analgesia will be provided by TCI Remifentanil. Following surgery, patients will be recovered by dedicated recovery nurses who will titrate intravenous morphine in the immediate postoperative period aiming to keep the NRS pain scores below 1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients will be receiving both interventions i.e. USG PECS blocks and wound infiltration anesthesia, with local anesthetic 0.25% levobupivacaine (active) and 0.9% Saline depending on the randomized group allocations. As such patients will be blinded.The anaesthetist and surgeon doing the interventions will both be blinded as to the pharmacological contents of the drug. This will be done as mentioned with pharmacy labelling the drugs as "PRE" used for USG pecs block and "POST" for wound infiltration. Also the observer, in this case the recovery nurse who will be titrating analgesia in the immediate postoperative period shall be blinded as to what group the patient belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group X (Active Comparator): PECS group
  USG PECS2 with Drug A (active) Wound infiltration with Drug P (placebo)
  Interventions: Procedure: USG PECS2 with Drug A (active); Procedure: Wound infiltration with Drug P (placebo)
- Group Y (Active Comparator): LA (local anaesthetic) infiltration group
  USG PECS2 with Drug P (placebo) Wound infiltration with Drug A (active)
  Interventions: Procedure: USG PECS2 with Drug P (placebo); Procedure: Wound infiltration with Drug A (active)

INTERVENTIONS:
Procedure: USG PECS2 with Drug A (active) — Ultrasound guided Pecs 2 blocks with 0.25% levobupivacaine
  Arms: Group X
Procedure: USG PECS2 with Drug P (placebo) — Ultrasound guided Pecs 2 blocks with placebo (0.9% saline)
  Arms: Group Y
Procedure: Wound infiltration with Drug P (placebo) — Wound infiltration at the end of surgery with Drug P (0.9% saline)
  Arms: Group X
Procedure: Wound infiltration with Drug A (active) — Wound infiltration at the end of surgery with 0.25% levobupivacaine
  Arms: Group Y

SUMMARY:
Breast cancer is the most common cancer for which women in the UK (United Kingdom) undergo surgery. A novel ultrasound guided regional anaesthetic technique called the 'Pecs 2' block has recently been described. This study compares ultrasound guided (USG) Pecs 2 block with local anaesthetic infiltration (LIA) for pain relief following breast cancer surgery.

DETAILED DESCRIPTION:
Breast cancer is the commonest cancer in UK for which women undergo surgery. Pain relief for breast surgery may be either opioid/morphine based or regional or local anesthetic technique based. Both have specific advantages and disadvantages. Regional anesthesia is known to suppress the stress response to surgery by blocking noxious afferent neural input into the central nervous system. Locoregional anesthetic techniques offer excellent pain relief without the disadvantages of morphine.These include thoracic epidural anesthesia, paravertebral block, intercostal blocks and local anesthetic infiltration of the wound. More recently, a novel ultrasound guided interfascial nerve block technique the 'Pecs block' was proposed by Blanco et al which provides an alternative method of providing postoperative analgesia for breast surgery.There is also evidence, albeit limited to support use of local anesthetic infiltration in breast surgery, which is widely used for analgesia.

Currently, there are no large randomised control trials to prove the safety and efficacy of ultrasound guided Pecs blocks in breast surgery. Also, wound infiltration with local anesthetic is practiced widely and to date, there has been no study comparing local anesthetic wound infiltration with USG pecs blocks.

On this background, we intend to perform a prospective randomised double blinded trial to evaluate the efficacy and safety of ultrasound guided Pecs blocks for breast surgery by comparing it local anesthetic wound infiltration.

This is a single-centre, prospective, double blinded randomised case control interventional study. The study plans to enroll 110 participants.

Patients will be randomly allocated to either group X or Y using computer generated numbers. Standard monitoring as per AAGBI (Association of anesthetists of Great Britain and Ireland) guidelines will be instituted as per clinical requirement. All patients will be anaesthetized using total intravenous anesthesia using TCI (target controlled infusions) of propofol and remifentanil. Intraoperatively, propofol and remifentanil infusions shall be titrated by the anesthetist to maintain adequate depth of anesthesia and analgesia.

Following induction of anesthesia and before surgical incision, all patients will receive USG modified Pecs 2 blocks as described by Blanco et al with 30 mls of pharmacy prepared Drug A (containing active drug that is 0.25% levobupivacaine) or Drug P (containing placebo 0.9% NaCl), labelled "PRE" (pre-surgery) respectively based on the group to which they are allocated.

At the end of surgery, the surgeon shall infiltrate the wound with 30 mls of Drug P or Drug A respectively, labelled "POST". (post-surgery)

The anesthetist and surgeon doing the interventions will both be blinded as to the pharmacological contents of the drug. This will be done as previously mentioned with pharmacy labelling the drugs as "PRE" used for USG pecs block and "POST" for wound infiltration.

Also the observer, in this case the recovery nurse who will be titrating analgesia in the immediate postoperative period shall be blinded as to what group the patient belongs to. Intraoperative analgesia will be provided by TCI remifentanil. It shall be supplemented in all patients with intravenous paracetamol and parecoxib as part of a multimodal analgesic technique. Following completion of surgery, the patients will be recovered by two dedicated recovery nurses. The nurses will titrate intravenous morphine in the immediate postoperative period aiming to keep the NRS (Numerical rating Scale) pain scores below 1.

Observations will be made in the intraoperative & postoperative period looking at relevant outcome measures. Patients shall be followed up at 1h, 6h and 24 hrs to collect primary outcome measures. Secondary outcomes will be collected by telephonic follow up at 6 months and 12 month intervals following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult female breast cancer patients
* Admitted to Craigavon Area Hospital
* Requiring and undergoing elective/urgent unilateral breast surgery as set out in the protocol

Exclusion Criteria:

* Patient allergic to local anaesthetic
* Any condition precluding safe use of USG pecs blocks e.g. Infection at site, anatomical abnormality etc.
* Preoperative chronic pain and or on pain medication over and above simple analgesics. Patients receiving any analgesia other than paracetamol, NSAIDS and codeine shall be excluded from the study.
* Bilateral breast surgery
* Consent declined

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only female participants
Enrollment: 110 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in Recovery | 24 hours
  A measure of total amount in milligrams of morphine required in recovery
Numeric Rating Scale (NRS) Pain scores | 24 hours
  Self reported pain scores between 0-10 (0- no pain; 10- severe pain, as bad as can be) in recovery

SECONDARY OUTCOMES:
PONV (Post operative nausea and vomiting) Impact Scale Score | 2 hours
  Measures Incidence and severity of postoperative nausea and vomiting before discharge from recovery
  Q1. Have you vomited or had dry retching?
  0 No
  1. Once
  2. Twice
  3. Three or more times Q2. Have you experienced a feeling of nausea (an unsettled feeling in the stomach and a slight urge to vomit) If yes, has your feeling of nausea interfered with activities of daily living, such as being able to get out of bed, being able to move about freely in bed, being able to eat normally, or eating and drinking?
  0 Not at all
  1. sometimes
  2. Often or most of the time
  3. All the time
  To calculate the PONV Impact Scale score, add the numerical responses to questions 1 and 2. A PONV Impact Scale score >5 defines clinically important PONV
S -LANNS (Self- administered Leeds Assessment of Neuropathic Symptoms and Signs) questionnaire for chronic post surgical pain | 1 year
  Incidence of chronic post surgical pain following unilateral breast and axillary surgery for breast cancer
Cancer recurrence or metastasis | 1 year
  Incidence of cancer recurrence or new metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Shiva K Arava, MD,FRCA,EDRA, Principal Investigator — Craigavon Area Hospital, SHSCT
Locations (1):
- Craigavon Area Hospital, Portadown, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonnema J, van Wersch AM, van Geel AN, Pruyn JF, Schmitz PI, Paul MA, Wiggers T. Medical and psychosocial effects of early discharge after surgery for breast cancer: randomised trial. BMJ. 1998 Apr 25;316(7140):1267-71. doi: 10.1136/bmj.316.7140.1267. PMID 9554895
- [Background] Bundred N, Maguire P, Reynolds J, Grimshaw J, Morris J, Thomson L, Barr L, Baildam A. Randomised controlled trial of effects of early discharge after surgery for breast cancer. BMJ. 1998 Nov 7;317(7168):1275-9. doi: 10.1136/bmj.317.7168.1275. PMID 9804712
- [Background] Purushotham AD, McLatchie E, Young D, George WD, Stallard S, Doughty J, Brown DC, Farish C, Walker A, Millar K, Murray G. Randomized clinical trial of no wound drains and early discharge in the treatment of women with breast cancer. Br J Surg. 2002 Mar;89(3):286-92. doi: 10.1046/j.0007-1323.2001.02031.x. PMID 11872051
- [Background] Bonnema J, van Wersch AM, van Geel AN, Pruyn JF, Schmitz PI, Uyl-de Groot CA, Wiggers T. Cost of care in a randomised trial of early hospital discharge after surgery for breast cancer. Eur J Cancer. 1998 Dec;34(13):2015-20. doi: 10.1016/s0959-8049(98)00258-5. PMID 10070303
- [Background] Exadaktylos AK, Buggy DJ, Moriarty DC, Mascha E, Sessler DI. Can anesthetic technique for primary breast cancer surgery affect recurrence or metastasis? Anesthesiology. 2006 Oct;105(4):660-4. doi: 10.1097/00000542-200610000-00008. PMID 17006061
- [Background] Sacerdote P, Bianchi M, Gaspani L, Manfredi B, Maucione A, Terno G, Ammatuna M, Panerai AE. The effects of tramadol and morphine on immune responses and pain after surgery in cancer patients. Anesth Analg. 2000 Jun;90(6):1411-4. doi: 10.1097/00000539-200006000-00028. PMID 10825330
- [Background] Yeager MP, Colacchio TA, Yu CT, Hildebrandt L, Howell AL, Weiss J, Guyre PM. Morphine inhibits spontaneous and cytokine-enhanced natural killer cell cytotoxicity in volunteers. Anesthesiology. 1995 Sep;83(3):500-8. doi: 10.1097/00000542-199509000-00008. PMID 7661350
- [Background] Naja MZ, Ziade MF, Lonnqvist PA. Nerve-stimulator guided paravertebral blockade vs. general anaesthesia for breast surgery: a prospective randomized trial. Eur J Anaesthesiol. 2003 Nov;20(11):897-903. doi: 10.1017/s0265021503001443. PMID 14649342
- [Background] Pusch F, Freitag H, Weinstabl C, Obwegeser R, Huber E, Wildling E. Single-injection paravertebral block compared to general anaesthesia in breast surgery. Acta Anaesthesiol Scand. 1999 Aug;43(7):770-4. doi: 10.1034/j.1399-6576.1999.430714.x. PMID 10456819
- [Background] Byager N, Hansen MS, Mathiesen O, Dahl JB. The analgesic effect of wound infiltration with local anaesthetics after breast surgery: a qualitative systematic review. Acta Anaesthesiol Scand. 2014 Apr;58(4):402-10. doi: 10.1111/aas.12287. PMID 24617619
- [Background] Campbell I, Cavanagh S, Creighton J, French R, Banerjee S, Kerr E, Shirley R. To infiltrate or not? Acute effects of local anaesthetic in breast surgery. ANZ J Surg. 2015 May;85(5):353-7. doi: 10.1111/ans.12541. Epub 2014 Apr 22. PMID 24754798
- [Background] Lynch EP, Welch KJ, Carabuena JM, Eberlein TJ. Thoracic epidural anesthesia improves outcome after breast surgery. Ann Surg. 1995 Nov;222(5):663-9. doi: 10.1097/00000658-199511000-00009. PMID 7487214
- [Background] Vila H Jr, Liu J, Kavasmaneck D. Paravertebral block: new benefits from an old procedure. Curr Opin Anaesthesiol. 2007 Aug;20(4):316-8. doi: 10.1097/ACO.0b013e328166780e. PMID 17620838
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Background] Bennett MI, Smith BH, Torrance N, Potter J. The S-LANSS score for identifying pain of predominantly neuropathic origin: validation for use in clinical and postal research. J Pain. 2005 Mar;6(3):149-58. doi: 10.1016/j.jpain.2004.11.007. PMID 15772908
- See also: Related Info — http://www.ons.gov.uk/ons/rel/vsob1/cancer-statistics-registrations--england--series-mb1-/index.html
- See also: Related Info — http://www.isdscotland.org/Health-Topics/Cancer/Publications/index.asp
- See also: Related Info — http://www.wales.nhs.uk/sites3/page.cfm?orgid=242&pid=59080